CLINICAL TRIAL: NCT02861703
Title: The Feasibility, Acceptability and Preliminary Effectiveness of an Online Lifestyle Intervention for Healthy Weight Management and Improved Quality of Life in Breast Cancer Survivors
Brief Title: Pilot Feasibility Study of an Online Lifestyle Intervention for Overweight Breast Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Canadian Breast Cancer Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CBCF-092014
Record Dates: First submitted 2015-12-11; First posted 2016-08-10 (Estimated); Last update posted 2018-12-21 (Actual); Status verified 2018-12

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Online lifestyle intervention (Experimental): A weekly psychosocial intervention ("Online Lifestyle Intervention") delivered in an online group format, to promote positive changes in physical (eating habits, physical activity) and mental health (body image, self-esteem, self-efficacy).
  Interventions: Behavioral: Online lifestyle intervention

INTERVENTIONS:
Behavioral: Online lifestyle intervention — Online, computer-mediated interactive group-based lifestyle intervention addressing thoughts, feelings, behaviours related to eating, physical activity, and other psychosocial issues related to breast cancer survivorship (e.g., mood, body image, existential issues, social support).

SUMMARY:
Obesity presents serious psychological and physical consequences for breast cancer survivors, including diminished quality of life, poorer prognosis and increased mortality. As such, there is a great need to develop strategies for these women to maintain optimal body weight. Diet and exercise have been shown to lead to successful weight loss among this population but these effects are seldom sustained, plausibly because these efforts alone overlook less obvious, but equally important, psychosocial factors that can interfere with prolonged progress. This study will implement a group-based intervention addressing diet and exercise along with other psychosocial issues related to survivorship such as depression, fatigue, body image and social support. Based on the growing popularity and benefits of computer-based health care, including convenience and anonymity, this intervention will also be offered online, representing the first of its kind. It is hypothesized that the intervention will be feasible to implement and acceptable to its participants. It is also hypothesized that the intervention will yield meaningful and sustained changes in body weight, body mass index, waist circumference (primary outcomes), as well as mental well-being, quality of life, and body image (secondary outcomes). This research has the ability to improve the long-term health of breast cancer survivors by incorporating psychosocial interventions into standard medical care practices and has the potential to increase accessibility of these services using online technology.

DETAILED DESCRIPTION:
Breast cancer (BC) is one of the most common types of cancer in Canadian women, and although the mortality rate is decreasing, there remain numerous challenges for survivorship. Among the most prevalent yet less commonly discussed post-treatment concerns, is substantial weight gain, with approximately 70% of women being overweight at diagnosis and additional weight gain often resulting from treatment. Obesity has serious psychological and physical implications for both pre- and post-menopausal BC survivors; in addition to compromising body image and QoL, it increases risk for recurrence and mortality. Specifically, increased fat results in greater production of estrogen, insulin, leptin and pro-inflammatory cytokines, and lesser production of sex hormone binding globulin, all of which have been linked to the promotion of BC and tumor growth. As such, the development of strategies for the promotion and maintenance of optimal body mass has become a primary focus for BC survivorship.

Trials of lifestyle interventions for this population are in their early stages and have primarily included modification of diet alone, exercise alone, or both. Results have been mixed, especially regarding the effects of dietary change alone but generally support the benefits of exercise and combined diet and exercise on weight loss and improved QoL in cancer survivors. However, despite indications that diet and exercise interventions lead to improvements in physical health and mental health, there remains a lack of consistent evidence that these gains are maintained long-term. As such, there is a need for more systematic follow-up of these interventions to determine their potential to produce enduring effects as well as for development and refinement of techniques that improve long-term weight management.

Beyond developing effective services, a direction for future research should include outreach to underserved populations. Rural BC survivors represent one group, in particular, with limited access to healthy lifestyle interventions, and who could benefit greatly from participation. Compared to their urban counterparts, these women are less likely to have timely diagnostic biopsies and receive optimal treatment, and are diagnosed later, at more advanced stages when prognosis is less favourable. They are also more likely to be obese, be less physically active, have poor eating habits, experience psychological distress, and have less access to mental health resources, placing them at heightened risk for weight gain. Researchers and health care providers have a responsibility to develop ways of redressing such health disparities and helping these particularly vulnerable women make lasting changes to their overall health and QoL.

Society's recent movement toward "eHealth", which refers to "the use of emerging information and communication technology, especially the Internet, to improve or enable health and health care", introduces an exciting opportunity to increase availability of health care to BC survivors. Numerous eHealth diet and exercise interventions have been evaluated using community samples and have generally yielded mixed findings along with recommendations for refinement of future programs and more rigorous evaluation. Only one online community intervention has been in group-format, and to the investigators knowledge, no online, group-based lifestyle intervention has yet been developed specifically for BC survivors. Given the potential for broader delivery of health care services via the Internet, research surrounding the value of computer-based lifestyle interventions is especially warranted.

Present Study

Firstly, while trials to date demonstrate that diet and exercise interventions lead to improvements in physical and mental health, there remains a lack of consistent evidence that these gains are maintained long-term. Arguably, programs that focus primarily on modifying nutrition and/or physical activity render only short-term effects because they fail to address more subtle, but ingrained, psychosocial factors that interfere with sustained progress. This project will develop and evaluate a group-based lifestyle intervention that incorporates diet and exercise strategies along with education of issues more broadly related to healthy lifestyle in the context of BC survivorship such as depression, fatigue, body image, and social support. The program will be developed by an interdisciplinary team of clinicians/researchers (oncologist, nurse, dietician, physiotherapist and senior psychologist), and grounded in Systems and Self-Determination Theory, which recognize one's motivation and self-efficacy as being the multi-determined product of interactions between personal, social, and environmental factors; as such, this program goes beyond behavioural diet and exercise modification by incorporating self-monitoring, motivational interviewing, professional knowledge, and peer feedback.

Secondly, despite growing evidence for the efficacy of interactive computer-based programs aimed at behaviour change and the associated advantages (e.g., convenience, accessibility, anonymity), there are no such interventions to support weight loss and sustained management for BC survivors. This project aims to fill this gap in health care by developing and evaluating the first online, group-based lifestyle intervention for BC survivors.

Objectives. The primary aim of this study is to evaluate the feasibility and acceptability of an online group-based lifestyle intervention for BC survivors. Qualitative data from the post-treatment interviews, and written responses from the treatment satisfaction survey were analyzed using thematic analysis to investigate this aim. A secondary aim is to evaluate the short- and longer-term effects of this healthy lifestyle intervention on participants' (1) physical (weight, BMI, waist circumference,) (2) behavioural (eating and physical activity habits) and (3) psychosocial well-being (quality of life, body image). This secondary aim was evaluated by comparing participants' scores on these measures prior to participating in the intervention, to their scores immediately following treatment, six months following treatment, and 12-months following treatment.

Primary aim hypotheses. It is hypothesized that this program is feasible to implement, as demonstrated by acceptable rates of attrition, homework completion and discussion board posting. It is also hypothesized that this program is acceptable, as demonstrated by satisfactory feedback obtained through a treatment satisfaction questionnaire and post-treatment interviews.

Secondary aim hypotheses. It is hypothesized that there will be a significant reduction in participants' weight, BMI, and waist circumference from pre-treatment to post-treatment, from pre-treatment to 6-months follow-up, and from pre-treatment to 12-months follow-up. It is hypothesized that there will be a significant improvement in participants' eating and physical activity habits from pre-treatment to post-treatment, from pre-treatment to 6-months follow-up, and from pre-treatment to 12-months follow-up. It is also hypothesized that there will be a significant improvement in participants' quality of life from pre-treatment to post-treatment, from pre-treatment to 6-months follow-up, and from pre-treatment to 12-months follow-up. Finally, it is hypothesized that there will be a significant improvement in participants' body image from pre-treatment to post-treatment, from pre-treatment to 6-months follow-up, and from pre-treatment to 12-months follow-up.

Method

This study will employ a single-arm pilot study, with repeated measures psychometric evaluation. Standardized measures will be completed at pre-treatment, post-treatment, and 6- and 12- months follow-up.

Recruitment

Participants will be accrued through the Louise Temerty Breast Center at Sunnybrook Health Sciences Centre (SHSC). The study will be advertised by staff and through brochures in the hospital and community-based organizations such as 'Willow Breast Cancer Support Canada', and via electronic brochures posted on websites commonly accessed by BC survivors. Interested women will contact the principal investigator, who will provide detailed information about the nature of the project, the study objectives and procedures, answer any questions the prospective participants have, and determine eligibility using the screening questionnaire.

Procedure

Participants will follow an individualized diet and exercise plan while participating in a 10-week online group, consisting of group discussion, educational videos, as well as homework completion and related feedback. Once screened, participants will be invited to SHSC to complete consent forms and baseline measures and a demographics questionnaire. They will be asked to complete these same measures immediately following completion of the intervention, as well as 6 and 12 months afterwards.

ELIGIBILITY:
Inclusion Criteria:

1. be 21 years or older
2. have been diagnosed with primary BC (stages I-III)
3. have completed active treatment within the previous 5 years
4. have a BMI above 25 or report a weight increase of 10 pounds or more post-treatment,
5. be available to participate in 10 consecutive weeks of the online program

7) be comfortable using and have access to a computer and secure Internet connection 8) can read and write in English.

Exclusion Criteria:

1. diagnosis of metastatic cancer
2. diagnosis of a mental health condition that would interfere with their own, or another group members' ability to benefit from the group (e.g., psychosis)
3. diagnosis of an additional medical condition that is not being successfully managed/treated
4. plans to undergo a medical procedure within the next year
5. plans to participate in another structured weight loss program or take weight loss medication within the next year.

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Change in Body Mass Index | Baseline, 6 months (mid-treatment), 12 months (post-treatment), 18 months (6-month follow-up), 24 months (12-month follow-up)
  Measured as a function of participants' weight (kg), divided by their height (squared metres)
Change in Waist Circumference | Baseline, 6 months (mid-treatment), 12 months (post-treatment), 18 months (6-month follow-up), 24 months (12-month follow-up)
  Measured as the difference across time points on participants' waist circumference in inches, using a nonelastic measuring tape at the widest part of hips.

SECONDARY OUTCOMES:
Change in Quality of Life | Baseline, 6 months (mid-treatment), 12 months (post-treatment), 18 months (6-month follow-up), 24 months (12-month follow-up)
  Measured as the difference across time points on participants' scores on the Functional Assessment of Cancer Therapy - For Patients with Breast Cancer (FACT-B)
Change in Subjective Health | Baseline, 6 months (mid-treatment), 12 months (post-treatment), 18 months (6-month follow-up), 24 months (12-month follow-up)
  Measured as the difference across time points on participants' scores on the Rand Health Survey--Short Form (SF-36)
Change in Life Satisfaction | Baseline, 6 months (mid-treatment), 12 months (post-treatment), 18 months (6-month follow-up), 24 months (12-month follow-up)
  Measured as the difference across time points on participants' scores on the Satisfaction with Life Scale (SWLS)
Change in Symptoms of Anxiety and Depression | Baseline, 6 months (mid-treatment), 12 months (post-treatment), 18 months (6-month follow-up), 24 months (12-month follow-up)
  Measured as the difference across time points on participants' scores on the Hospital Anxiety and Depression Scale (HADS)
Change in Body Image | Baseline, 6 months (mid-treatment), 12 months (post-treatment), 18 months (6-month follow-up), 24 months (12-month follow-up)
  Measured as the difference across time points on participants' scores on the Body Image Scale (BIS)
Change in Objectified Body Consciousness | Baseline, 6 months (mid-treatment), 12 months (post-treatment), 18 months (6-month follow-up), 24 months (12-month follow-up)
  Measured as the difference across time points on participants' scores on the Objectified Body Consciousness Scale (OBCS)
Change in Dietary Intake | Baseline, 6 months (mid-treatment), 12 months (post-treatment), 18 months (6-month follow-up), 24 months (12-month follow-up)
  Measured as the difference across time points on participants' scores on the Automated Self-administered 24-hour Dietary Recall (ASA24)
Change in 'Intuitive Eating' Habits | Baseline, 6 months (mid-treatment), 12 months (post-treatment), 18 months (6-month follow-up), 24 months (12-month follow-up)
  Measured as the difference across time points on participants' scores on the Intuitive Eating Scale-2 (IES-2)
Change in Exercise Habits | Baseline, 6 months (mid-treatment), 12 months (post-treatment), 18 months (6-month follow-up), 24 months (12-month follow-up)
  Measured as the difference across time points on participants' scores on the Godin Leisure-Time Exercise Questionnaire
Change in Self-Efficacy | Baseline, 6 months (mid-treatment), 12 months (post-treatment), 18 months (6-month follow-up), 24 months (12-month follow-up)
  Measured as the difference across time points on participants' scores on the Nutrition and Physical Exercise Self-Efficacy Scale

CONTACTS AND LOCATIONS:
Overall Officials: Karen Fergus, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada